CLINICAL TRIAL: NCT03293134
Title: Clinical and Molecular Characterization of Cerebral Proliferative Vasculopathy
Acronym: VPCA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI11031
Record Dates: First submitted 2017-05-02; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-03

CONDITIONS: Proliferative Vasculopathy
Keywords: Fowler syndrome
MeSH Terms: conditions — Fowler Christmas Chapple syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood, cells cultivated, extracted DNA and fetal tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As principal objective, the study aims to:

1. Describe the spectrum and evaluate the frequency of angiodysplasia of the nevrax;
2. Establish the physiopathological basis of Fowler's syndrome;
3. Identify FLVCR2 partners and the signaling pathways involved;
4. Test new candidate genes: GPR124 and possible partners of FLVCR2.

As second objective, the study aims to:

* perform phenotype / genotype correlation if necessary;
* and propose a prenatal diagnosis in families with identified mutations.

ELIGIBILITY:
Inclusion Criteria:

* Angiodysplasia restricted to central nervous system with or without glomerular vasculopathy.
* Informed consent signed.

Exclusion Criteria:

* Vascular malformations not confined to the nevrax.
* No signature of consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intrauterine fetal death and those from termination of pregnancy for fetal abnormality.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2015-03-09 (Actual); Study Completion 2016-10-06 (Actual)

PRIMARY OUTCOMES:
Morphological analysis | throughout the study: 36 months
  Morphological analysis : characterisation of cellular lesions by immunolabelling with endothelial markers such as CD34 and CD31, pericytic markers (smooth muscle actin and proteoglycan NG2) and astrocytic markers (GFAP)

SECONDARY OUTCOMES:
Identification of novel disease | throughout the study: 36 months
  Identification of novel disease causing genes in addition to FLVCR2 by whole exome sequencing.
  Fetus with clinical VPCA and no FLVCR2 mutation found by Sanger sequencing, will be studied by whole exome sequencing in order to find mutation in other genes that could explain the phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Attié-Bitach, MD, PhD, Principal Investigator — Hôpital Necker Enfants Malades, APHP
Locations (1):
- Hôpital Necker Enfants Malades, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomas S, Encha-Razavi F, Devisme L, Etchevers H, Bessieres-Grattagliano B, Goudefroye G, Elkhartoufi N, Pateau E, Ichkou A, Bonniere M, Marcorelle P, Parent P, Manouvrier S, Holder M, Laquerriere A, Loeuillet L, Roume J, Martinovic J, Mougou-Zerelli S, Gonzales M, Meyer V, Wessner M, Feysot CB, Nitschke P, Leticee N, Munnich A, Lyonnet S, Wookey P, Gyapay G, Foliguet B, Vekemans M, Attie-Bitach T. High-throughput sequencing of a 4.1 Mb linkage interval reveals FLVCR2 deletions and mutations in lethal cerebral vasculopathy. Hum Mutat. 2010 Oct;31(10):1134-41. doi: 10.1002/humu.21329. PMID 20690116